CLINICAL TRIAL: NCT03399162
Title: PRehabilitiation in Elective Frail and Elderly Cardiac Surgery PaTients (PREFECT): Assessing the Impact of a Personalized Prehabilitation Program Before Cardiac Surgery on Frailty and Clinical Outcomes
Brief Title: PRehabilitiation in Elective Frail and Elderly Cardiac Surgery PaTients
Acronym: PREFECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a reduction in surgical wait times, there was insufficient time to complete the intervention prior to surgery.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20170698
Record Dates: First submitted 2017-09-20; First posted 2018-01-16 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREHAB Group (Experimental): Patients in this arm will receive the usual standard of care prior to surgery, which includes a PREHAB workshop; consultations with a surgeon, anaesthesiologist, and nurse; referrals to diabetes counselling and/or smoking cessation, as appropriate; and the usual diagnostic work-up.
  Patients in this group will also complete an 8-week PREHAB exercise program, with weekly exercise classes and a list of exercises to complete at home.
  Interventions: Behavioral: PREHAB Workshop; Behavioral: PREHAB Exercise Program
- Standard of care group (Active Comparator): Patients in this arm will receive the usual standard of care prior to surgery, which includes a PREHAB workshop; consultations with a surgeon, anaesthesiologist, and nurse; referrals to diabetes counselling and/or smoking cessation, as appropriate; and the usual diagnostic work-up.
  Interventions: Behavioral: PREHAB Workshop

INTERVENTIONS:
Behavioral: PREHAB Workshop — PREHAB workshop/education session in the Prevention and Rehabilitation Centre regarding nursing, nutrition, physiotherapy, psychology, and diabetes.
Behavioral: PREHAB Exercise Program — An 8-week program that consists of: (1) 2x/week 60-minute supervised exercise sessions; and (2) 3x/week 30-minute home-based exercise sessions.
  Arms: PREHAB Group

SUMMARY:
Older and more frail adults are more often being referred for cardiac surgery. These patients are often in suboptimal health, and may be physically frail, malnourished, and have other conditions, such as diabetes, that complicate their recovery. Research suggests that a rehabilitation program prior to surgery may help improve participants' health and improve their fitness for surgery. Currently, a pre-operative rehabilitation workshop is offered at the University of Ottawa Heart Institute, but this interventional, randomized study will investigate whether a more comprehensive pre-operative regime, including structured weekly exercise program, is more effective at improving health prior to surgery. Patients will be randomized to either the control group (pre-operative rehabilitation workshop ONLY) or the treatment group (pre-operative rehabilitation workshop plus exercise regime). This regime will attempt to improve patients' overall health, including their physical fitness and nutritional status. The effectiveness of this regime will be evaluated by comparing patients' physical function, questionnaires (diet, quality of life, stress) and serum biomarkers from baseline to pre-surgery to post-surgery. The Investigators hypothesize that patients that complete the pre-operative rehabilitation program will improve their health prior to surgery, and that this may result in shorter length of hospitalization and fewer complications after surgery. The study will take place over two years, with each patient's participation lasting about 3 months.

DETAILED DESCRIPTION:
Frailty is a common syndrome among older adults, defined as a "clinically recognizable state of increased vulnerability resulting from aging-associated decline in reserve and function". Fried defined frailty as meeting three out of the five criteria: low grip strength, low energy, slowed walking speed, low physical activity, and/or unintentional weight loss. Clinicians are currently challenged with a rising prevalence of elderly and frail patients presenting for major cardiac surgery. Such patients typically present with a greater comorbidity burden and are more likely to be malnourished, physically deconditioned, and to exhibit decreased physiological adaptation to stress. Frail cardiac surgical patients are, unsurprisingly, at increased risk for major adverse cardiac and cerebrovascular events, short- and longer-term mortality, and increased length of hospital of stay. Clinicians may also struggle to quantify the peri-operative risk of morbidity and mortality among these individuals, since tools such as the Society of Thoracic Surgeons (STS) risk assessment are not designed to comprehensively assess the complex interaction between various risk factors seen in the frail patient.

Cardiovascular rehabilitation (CR) programs are integral to managing patients with cardiovascular disease. Such programs include health behaviour change, and cardiovascular risk factor management (e.g. moderate-to-vigorous-intensity continuous exercise training [MICE], healthy eating, smoking cessation, stress management, and psychological services). The benefits of MICE for patients with cardiovascular disease include improvements in exercise tolerance, muscular strength, cardiovascular health and reduced hospitalizations. MICE is, therefore, able to improve several facets of physical dysfunction, and forms major therapeutic interventions for functional capacity and frailty. Improvements in nutritional status have been observed in patients with cardiovascular disease(CVD) participating in CR, and exercise training and stress management have been shown to reduce distress in CVD patients.

Emerging evidence indicates that CR before cardiac surgery (i.e. prehabilitation [PREHAB]) may improve clinical outcomes. Sawatzky et al. showed that a 12-week PREHAB program consisting of two structured exercise training sessions per week and 12 education sessions concerning cardiovascular risk factor management, exercise, stress, diet, and medication use in patients awaiting coronary artery bypass grafting (CABG) was feasible and significantly improved functional capacity.

Elderly and frail patients are increasingly presenting for cardiac surgery, and these individuals must be carefully optimized pre-operatively to increase the likelihood of their recovery and return to a reasonable quality of life. A personalized PREHAB program that targets and ameliorates the elements of frailty, including low functional capacity, poor nutrition, and stress, offers the best chance of mitigating frailty and its associated risk factors in a way that is feasible, patient-centred, and translatable to other cardiovascular centres. This project will use objective measures, including tests of functional capacity, validated questionnaires, and biomarker analysis, to better quantify the subjective diagnosis of frailty in our patients, and will implement a novel personalized PREHAB program with integrated on-site and home-based exercise sessions, in an attempt to mitigate the frailty and other risk factors that impact patients in the peri-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Patients able to provide informed consent
* Patients undergoing elective cardiac surgery for either CABG, valve, or CABG + valve
* Patients who have an estimated wait time of at least 10 weeks.
* Patients who are either ≥65 years of age or classified as frail using Fried Frailty criteria or scoring at least 3 on the Clinical Frailty Scale

Exclusion Criteria:

* Patients with current or recent unstable cardiac disease, defined as and of the following:
* CCS class IV angina,
* NYHA Class III or IV heart failure,
* Critical left main disease,
* hospitalization for arrhythmia within the last month
* Dynamic ventricular outflow obstruction
* Symptomatic exercise-induced arrhythmia
* Patients who are cognitively, geographically or physically unable to complete the PREHAB sessions
* Patients who, in the opinion of either their treating physician or the study investigators, should not participate in a pre-operative rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | Change between baseline and 8 weeks (+/- 1 week)
  The primary outcome, functional capacity, will be measured using the 6-minute walk test.

SECONDARY OUTCOMES:
Frailty (Fried criteria) | Compared between baseline, 8 weeks (+/- 1 week), and 4 weeks after surgery (+/- 2 weeks)
  Measured using the Fried frailty score (presence of 3 of the 5 symptoms of frailty)
Frailty (clinical score) | Compared between baseline, 8 weeks (+/- 1 week), and 4 weeks after surgery (+/- 2 weeks)
  Measured using the Clinical Frailty Scale (9 point clinical assessment)
Short Form - 36 | Compared between baseline, 8 weeks (+/- 1 week), and 4 weeks after surgery (+/- 2 weeks)
  Measured using the SF-36 Quality of Life questionnaire
Depression | Compared between baseline, 8 weeks (+/- 1 week), and 4 weeks after surgery (+/- 2 weeks)
  Measured using the BDI-II
Anxiety | Compared between baseline, 8 weeks (+/- 1 week), and 4 weeks after surgery (+/- 2 weeks)
  Measured using the BAI
Dietary habits | Compared between baseline, 8 weeks (+/- 1 week), and 4 weeks after surgery (+/- 2 weeks)
  Measured using the Block food frequency questionnaire
Exercise adherence | Compared between baseline and 8 weeks (+/- 1 week)
  Measured using a pedometer
Clinical and cardiovascular outcomes | In the 6 weeks after surgery
  A composite endpoint that will look at the rates of occurrence of major cardiovascular and cerebrovascular outcomes (i.e. death, myocardial infarction, cardiac arrest, stroke) and length of hospitalization.

OTHER OUTCOMES:
Biomarkers | Compared between baseline and 8 weeks (+/- 1 week)
  An exploratory outcome where we will examine a panel of biomarkers to determine the biomarker profile of frail and elderly patients referred for cardiac surgery, and to observe what changes, if any, occur after the PREHAB intervention. The biomarker panel includes markers of cardiovascular health and risk (NT-pro BNP, cholesterol, homocysteine), nutritional status (albumin, prealbumin, trasnferrin receptor, 25-hydroxy-vitamin D), inflammation (interleukin 6, selenium, high sensitivity CRP, sRAGE), renal function (creatinine, cystatin C), liver function (AST, ALT), and overall health (CBC, adiponectin, dehydroepiandrosterone sulfate, sex hormone-binding globulin, insulin-like growth factor).

CONTACTS AND LOCATIONS:
Overall Officials: Juan B Grau Alvaro, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Louise Sun, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Jennifer Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Afilalo J, Mottillo S, Eisenberg MJ, Alexander KP, Noiseux N, Perrault LP, Morin JF, Langlois Y, Ohayon SM, Monette J, Boivin JF, Shahian DM, Bergman H. Addition of frailty and disability to cardiac surgery risk scores identifies elderly patients at high risk of mortality or major morbidity. Circ Cardiovasc Qual Outcomes. 2012 Mar 1;5(2):222-8. doi: 10.1161/CIRCOUTCOMES.111.963157. Epub 2012 Mar 6. PMID 22396586